CLINICAL TRIAL: NCT05809362
Title: Validation of a Photoplethysmography-Based Algorithm for Detection of Atrial Fibrillation Via a Wearable Device - WHOOP Abnormal Rhythm Notification
Brief Title: WHOOP Abnormal Rhythm Notification
Acronym: WARN
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Whoop Inc. (Industry); ZS Associates, Inc. (Unknown)
Responsible Party: Principal Investigator, Francis P. Wilson, Associate Professor of Medicine, Yale University
Other Study IDs: 2000031382
Record Dates: First submitted 2023-03-29; First posted 2023-04-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Wearable device
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Atrial Fibrillation: Subjects with known diagnosis of atrial fibrillation (persistent or paroxysmal) documented in the medical record.
  Interventions: Device: WHOOP 4.0 Strap; Device: BioTel ePatch
- No atrial fibrillation: Subjects with no known diagnosis of atrial fibrillation as documented in the medical record.
  Interventions: Device: WHOOP 4.0 Strap; Device: BioTel ePatch

INTERVENTIONS:
Device: WHOOP 4.0 Strap — Subjects will receive both the WHOOP 4.0 Strap and the BioTel ePatch and will continuously wear each for one week. Data will be collected and analyzed by the study team upon return of the both devices from the subject.
Device: BioTel ePatch — Subjects will receive both the WHOOP 4.0 Strap and the BioTel ePatch and will continuously wear each for one week. Data will be collected and analyzed by the study team upon return of the both devices from the subject.

SUMMARY:
The purpose of this protocol is to assess the sensitivity and specificity of a photoplethysmography (PPG)-based algorithm for the detection of atrial fibrillation as compared to a gold-standard assessment (wearable ECG patch) among a population of individuals with known atrial fibrillation and without known atrial fibrillation over a 7-day study period.

DETAILED DESCRIPTION:
Atrial fibrillation (Afib) is the most common cardiac arrhythmia in the United States, affecting up to one in four individuals across the lifespan, and is associated with substantial morbidity and mortality. Fifteen percent of strokes in the United States are attributable to Afib, and nearly 20% of these occur in individuals with no prior Afib history. Because Afib is often paroxysmal, one-time screening is unlikely to capture those at risk. Thus, there has been an increasing interest in leveraging monitoring for Afib via wearable devices, which provide a novel method to detect Afib and determine the burden of Afib in the general population. Devices such as the WHOOP 4.0 strap use advanced sensors to detect pulse rate and other physiologic metrics in real-time. Given the high degree of pulse-rate variability in Afib, it is clear that algorithms evaluating data from these devices may be able to detect asymptomatic Afib. However, the sensitivity and specificity of the algorithm operating on data from the WHOOP 4.0 strap have not been formally evaluated in a clinical setting.

The WHOOP strap measures changes in blood flow via photoplethysmography (PPG), from which timing between successive heartbeats ("beat-to-beat intervals") is measured. While normal sinus rhythm tends to display beat-to-beat intervals of similar magnitude, those of cardiac arrythmias are characterized by higher variability and may follow particular patterns.

The primary objective of this study is to assess the sensitivity and specificity of the WHOOP Strap ANF 1.0 classification algorithm for the detection of Afib as compared to a gold-standard assessment (one-week ECG patch monitoring using the BioTel ePatch).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 22 years
* Known diagnosis of atrial fibrillation OR no history of arrhythmia as documented in the patient medical record
* Seen in a Yale New Haven Hospital-associated Primary Care or Cardiology Clinic
* Cell phone (IOS 15.0 or greater or Android 10 or greater) with an active data plan and willing to install the WHOOP Mobile Application software
* Full-time US resident
* Able to read, understand, and provide written informed consent in English
* Willing and able to participate in the study procedures as described in the consent form
* Able to communicate effectively with and follow instructions from the study staff

Exclusion Criteria:

* Pre-existing WHOOP user with active account
* Has implantable cardiac device (e.g., pacemaker, ICD, LVAD)
* Solid organ transplant
* Sensitivity or allergy to ECG patch or skin glue
* Unwilling to wear WHOOP 4.0 strap for one week
* Unwilling to wear BioTel (ECG patch) ePatch for one week
* WHOOP strap should be the only wearable on the arm. Individuals unwilling to adhere to the proper usage of the WHOOP strap will be excluded.
* Unwilling to install the WHOOP Mobile Application software
* Unable to provide informed consent
* Non-English speaking (as the WHOOP Mobile Application software is English only)
* Known sensitivity to medical adhesives, isopropyl alcohol, watch bands, or electrocardiogram (ECG) electrodes including known allergy or sensitivity to polyamide, polyester, or elastane bands primarily used in wrist worn fitness devices
* Symptomatic (or active) allergic skin reactions
* Significant tremor that prevents the subject from being able to hold still.
* Acute myocardial infarction (MI) within 90 days of screening or other cardiovascular disease that, in the opinion of the investigator, increases the risk to the subject or renders data uninterpretable.
* Pregnant women: Women who report being pregnant at the time of study participation.
* Subjects taking rhythm control drugs including amiodarone, dronedarone, dofetilide, sotalol, flecainide, ibutilide, lidocaine, procainamide, propafenone, quinidine, tocainide.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include adults seen in primary care and cardiology clinics associated with a single health system. The prospective cohort will comprise three distinct populations - individuals with a known history of persistent atrial fibrillation, individuals with paroxysmal atrial fibrillation, and individuals without a history of cardiac arrhythmia of any kind.
Sampling Method: Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the PPG-based WHOOP ANF algorithm for detection of atrial fibrillation | 7 days of continuous wear of the WHOOP 4.0 Strap and BioTel ePatch immediately post enrollment
  Sensitivity is defined as the True Positives/(True Positives + False Negatives). A "true" atrial fibrillation reading will have an ECG patch reading consistent with sustained atrial fibrillation for at least 5 continuous minutes. A WHOOP ANF diagnosis of atrial fibrillation is defined as "atrial fibrillations" being detected using the internal algorithm. A true positive is defined as the count of individuals who have at least 1 window labelled as Afib by WHOOP ANF and which has 5+ minutes of continuous Afib as determined by the BioTel recording and confirmed by tachogram adjudication. A false negative is defined as individuals who do not have any windows labelled by WHOOP-ANF as having Afib but at least one window has 5+ minutes of continuous Afib as determined by the BioTel recording.
Specificity of the PPG-based WHOOP ANF algorithm for detection of atrial fibrillation | 7 days of continuous wear of the WHOOP 4.0 Strap and BioTel ePatch immediately post enrollment
  Specificity is defined as the True Negatives/(True Negatives + False Positives). A "true" atrial fibrillation reading will have an ECG patch reading consistent with sustained atrial fibrillation for at least 5 continuous minutes. A WHOOP ANF diagnosis of atrial fibrillation is defined as "atrial fibrillations" being detected using the internal algorithm. A true negative is defined as the count of individuals who do not have any windows labelled by WHOOP ANF as having Afib and none of these windows contain 5+ minutes of continuous Afib as determined by the BioTel recording. A false positive is defined as individuals who have windows labelled as Afib by WHOOP ANF but none of these windows contain 5 minutes or greater of continuous Afib as determined by BioTel recording or have 5+ minutes of continuous Afib as determined by BioTel recording but none can be verified by tachogram adjudication.

SECONDARY OUTCOMES:
Concordance between WHOOP ANF and BioTel ePatch via epoch assessment | 7 days of continuous wear of the WHOOP 4.0 Strap and BioTel ePatch immediately post enrollment
  Comparison of each epoch by both WHOOP ANF and the BioTel ePatch for concordance using the following definitions: True Positive: An epoch detected by WHOOP ANF as "atrial fibrillation" that has >=5 mins of AFib as detected by the ECG patch. True Negative: An epoch that is NOT labelled as "atrial fibrillation" by the WHOOP ANF and has < 5 mins of AFib as detected by the ECG patch. Specificity of the algorithm on the epoch level: True Negative/(True Negatives + False Positives). Sensitivity of the algorithm on the epoch level: True Positives / (True Positives + False Negatives). Positive predictive value of the algorithm on the epoch level: True Positives / (True Positives + False Positives). Negative predictive value of the algorithm on the epoch level: True Negatives / (True Negatives + False Negatives).

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Wilson, MD MSCE, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar S, Weinstein J, Melchinger HC, Smith A, Capodilupo E, Akar JG, Garg K, O'Connor KD, Staunton MK, Martin M, Akhlaghi N, Edeh O, Perez S, Lee V, Lee KAV, Wilson FP. Observational study protocol for an arrhythmia notification feature. BMJ Open. 2024 Jun 3;14(6):e075110. doi: 10.1136/bmjopen-2023-075110. PMID 38830741